CLINICAL TRIAL: NCT03317925
Title: Renal Transplant Injury and the Renin-Angiotensin System in Kids (RETASK)
Acronym: RETASK
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 00046001
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Renal Transplant; Renin-Angiotensin System; Rejection Acute Renal; Rejection Chronic Renal; Rejection of Renal Transplant
Keywords: Pediatric Renal Transplant; Renal Allograft; Angiotensin II; Angiotensin-(1-7); ACE; ACE2
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — De-identified urine and plasma specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Renal Transplantation — Kidney transplantation and biomarkers that can identify injury after transplant.

SUMMARY:
In pediatric kidney transplant patients, rejection, medication toxicity and ischemia cause early and chronic renal allograft injury, which reduces graft lifespan and patient survival. Early detection of injury would facilitate prevention and treatment. The gold standard surveillance biopsy has limitations including delayed discovery of injury. No noninvasive test identifies graft injury before it is clinically apparent. This project's goal is to develop a novel early marker of subclinical graft injury to facilitate prompt recognition and treatment.

DETAILED DESCRIPTION:
Kidney damage activates the traditional renin-angiotensin (Ang) system (RAS), characterized by Ang-converting enzyme (ACE)/Ang II/Ang II type 1 receptor. The Ang-converting enzyme 2 (ACE2)/Ang-(1-7)/Mas pathway counteracts this damage. The balance, or ratio, between levels of the ACE/Ang II and ACE2/Ang-(1-7) pathways may be clinically important because Ang-(1-7) counteracts Ang II-mediated injury. An increase in ACE and Ang II expression and a decrease in ACE2 and Ang-(1-7) expression on tubular cells may promote renal injury. Tubular damage may increase urinary loss of protective ACE2 and Ang-(1-7), propagating renal damage by allowing ACE and Ang II to stimulate inflammation and fibrosis unopposed. The investigators hypothesis is that a shift in the urinary ACE-to-ACE2 and Ang II-to-Ang-(1-7) ratios towards ACE2 and Ang-(1-7) predicts acute graft injury diagnosed on renal biopsy and predicts chronic graft damage on renal biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 - 20 years
* Actively listed on the transplant list at Lucile Packard Children's Hospital at Stanford and received a renal transplant during the study enrollment period

Exclusion Criteria:

* Transplanted at a center other than Lucile Packard Children's Hospital at Stanford

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is an observational study with a convenience sample of patients recruited from Lucile Packard Children's Hospital kidney transplant evaluation clinic.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Acute graft injury | Within six months after kidney transplant
  Renal biopsy-confirmed acute renal allograft injury as determined by a pathologist (binary yes or no)

SECONDARY OUTCOMES:
Chronic graft damage | Six months after kidney transplant
  Renal biopsy-confirmed chronic renal allograft damage as determined by a quantitative fibrosis pathology stain (percent fibrosis from 0 to 100%)
Renal function | Within six months after kidney transplant
  Glomerular filtration rate by the Schwartz equation (mL/min/1.73 m^2)
Proteinuria | Within six months after kidney transplant
  Urine protein-to-creatinine ratio above 0.2 mg/mg creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M South, MD MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furness PN, Taub N, Assmann KJ, Banfi G, Cosyns JP, Dorman AM, Hill CM, Kapper SK, Waldherr R, Laurinavicius A, Marcussen N, Martins AP, Nogueira M, Regele H, Seron D, Carrera M, Sund S, Taskinen EI, Paavonen T, Tihomirova T, Rosenthal R. International variation in histologic grading is large, and persistent feedback does not improve reproducibility. Am J Surg Pathol. 2003 Jun;27(6):805-10. doi: 10.1097/00000478-200306000-00012. PMID 12766585
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345
- [Background] Halawa A. The early diagnosis of acute renal graft dysfunction: a challenge we face. The role of novel biomarkers. Ann Transplant. 2011 Jan-Mar;16(1):90-8. PMID 21436782
- [Background] Hall IE, Yarlagadda SG, Coca SG, Wang Z, Doshi M, Devarajan P, Han WK, Marcus RJ, Parikh CR. IL-18 and urinary NGAL predict dialysis and graft recovery after kidney transplantation. J Am Soc Nephrol. 2010 Jan;21(1):189-97. doi: 10.1681/ASN.2009030264. Epub 2009 Sep 17. PMID 19762491
- [Background] Schaub S, Mayr M, Honger G, Bestland J, Steiger J, Regeniter A, Mihatsch MJ, Wilkins JA, Rush D, Nickerson P. Detection of subclinical tubular injury after renal transplantation: comparison of urine protein analysis with allograft histopathology. Transplantation. 2007 Jul 15;84(1):104-12. doi: 10.1097/01.tp.0000268808.39401.e8. PMID 17627245
- [Background] Ruster C, Wolf G. Renin-angiotensin-aldosterone system and progression of renal disease. J Am Soc Nephrol. 2006 Nov;17(11):2985-91. doi: 10.1681/ASN.2006040356. Epub 2006 Oct 11. PMID 17035613
- [Background] Iwai M, Horiuchi M. Devil and angel in the renin-angiotensin system: ACE-angiotensin II-AT1 receptor axis vs. ACE2-angiotensin-(1-7)-Mas receptor axis. Hypertens Res. 2009 Jul;32(7):533-6. doi: 10.1038/hr.2009.74. Epub 2009 May 22. PMID 19461648
- [Background] Ferrario CM. ACE2: more of Ang-(1-7) or less Ang II? Curr Opin Nephrol Hypertens. 2011 Jan;20(1):1-6. doi: 10.1097/MNH.0b013e3283406f57. PMID 21045683
- [Background] Santos RA, Ferreira AJ, Pinheiro SV, Sampaio WO, Touyz R, Campagnole-Santos MJ. Angiotensin-(1-7) and its receptor as a potential targets for new cardiovascular drugs. Expert Opin Investig Drugs. 2005 Aug;14(8):1019-31. doi: 10.1517/13543784.14.8.1019. PMID 16050794
- [Background] Santos RA, Ferreira AJ, Simoes E Silva AC. Recent advances in the angiotensin-converting enzyme 2-angiotensin(1-7)-Mas axis. Exp Physiol. 2008 May;93(5):519-27. doi: 10.1113/expphysiol.2008.042002. Epub 2008 Feb 29. PMID 18310257
- [Background] Dilauro M, Burns KD. Angiotensin-(1-7) and its effects in the kidney. ScientificWorldJournal. 2009 Jun 30;9:522-35. doi: 10.1100/tsw.2009.70. PMID 19578709
- [Background] Heringer-Walther S, Eckert K, Schumacher SM, Uharek L, Wulf-Goldenberg A, Gembardt F, Fichtner I, Schultheiss HP, Rodgers K, Walther T. Angiotensin-(1-7) stimulates hematopoietic progenitor cells in vitro and in vivo. Haematologica. 2009 Jun;94(6):857-60. doi: 10.3324/haematol.2008.000034. Epub 2009 Apr 18. PMID 19377080
- [Background] Geara AS, Azzi J, Jurewicz M, Abdi R. The renin-angiotensin system: an old, newly discovered player in immunoregulation. Transplant Rev (Orlando). 2009 Jul;23(3):151-8. doi: 10.1016/j.trre.2009.04.002. PMID 19539879
- [Background] Miyake-Ogawa C, Miyazaki M, Abe K, Harada T, Ozono Y, Sakai H, Koji T, Kohno S. Tissue-specific expression of renin-angiotensin system components in IgA nephropathy. Am J Nephrol. 2005 Jan-Feb;25(1):1-12. doi: 10.1159/000083224. Epub 2005 Jan 7. PMID 15644622
- [Background] Jurewicz M, McDermott DH, Sechler JM, Tinckam K, Takakura A, Carpenter CB, Milford E, Abdi R. Human T and natural killer cells possess a functional renin-angiotensin system: further mechanisms of angiotensin II-induced inflammation. J Am Soc Nephrol. 2007 Apr;18(4):1093-102. doi: 10.1681/ASN.2006070707. Epub 2007 Feb 28. PMID 17329576
- [Background] Su Z, Zimpelmann J, Burns KD. Angiotensin-(1-7) inhibits angiotensin II-stimulated phosphorylation of MAP kinases in proximal tubular cells. Kidney Int. 2006 Jun;69(12):2212-8. doi: 10.1038/sj.ki.5001509. Epub 2006 May 3. PMID 16672906
- [Background] Moon JY. ACE2 and Angiotensin-(1-7) in Hypertensive Renal Disease. Electrolyte Blood Press. 2011 Dec;9(2):41-4. doi: 10.5049/EBP.2011.9.2.41. Epub 2011 Dec 31. PMID 22438854
- [Background] Ahmed AK, El Nahas AM, Johnson TS. Changes in matrix metalloproteinases and their inhibitors in kidney transplant recipients. Exp Clin Transplant. 2012 Aug;10(4):332-43. doi: 10.6002/ect.2012.0013. PMID 22845765
- [Background] Castoldi G, di Gioia CR, Travaglini C, Busca G, Redaelli S, Bombardi C, Stella A. Angiotensin II increases tissue-specific inhibitor of metalloproteinase-2 expression in rat aortic smooth muscle cells in vivo: evidence of a pressure-independent effect. Clin Exp Pharmacol Physiol. 2007 Mar;34(3):205-9. doi: 10.1111/j.1440-1681.2007.04573.x. PMID 17250640
- [Background] Mazanowska O, Kaminska D, Krajewska M, Zabinska M, Kopec W, Boratynska M, Chudoba P, Patrzalek D, Klinger M. Imbalance of metallaproteinase/tissue inhibitors of metalloproteinase system in renal transplant recipients with chronic allograft injury. Transplant Proc. 2011 Oct;43(8):3000-3. doi: 10.1016/j.transproceed.2011.08.012. PMID 21996210
- [Background] Ling XB, Sigdel TK, Lau K, Ying L, Lau I, Schilling J, Sarwal MM. Integrative urinary peptidomics in renal transplantation identifies biomarkers for acute rejection. J Am Soc Nephrol. 2010 Apr;21(4):646-53. doi: 10.1681/ASN.2009080876. Epub 2010 Feb 11. PMID 20150539
- [Background] Lutz J, Yao Y, Song E, Antus B, Hamar P, Liu S, Heemann U. Inhibition of matrix metalloproteinases during chronic allograft nephropathy in rats. Transplantation. 2005 Mar 27;79(6):655-61. doi: 10.1097/01.tp.0000151644.85832.b5. PMID 15785371
- [Background] Pan CH, Wen CH, Lin CS. Interplay of angiotensin II and angiotensin(1-7) in the regulation of matrix metalloproteinases of human cardiocytes. Exp Physiol. 2008 May;93(5):599-612. doi: 10.1113/expphysiol.2007.041830. Epub 2008 Feb 22. PMID 18296491
- [Background] Clark MA, Tallant EA, Diz DI. Downregulation of the AT1A receptor by pharmacologic concentrations of Angiotensin-(1-7). J Cardiovasc Pharmacol. 2001 Apr;37(4):437-48. doi: 10.1097/00005344-200104000-00011. PMID 11300657
- [Background] Brosnihan KB, Neves LA, Joyner J, Averill DB, Chappell MC, Sarao R, Penninger J, Ferrario CM. Enhanced renal immunocytochemical expression of ANG-(1-7) and ACE2 during pregnancy. Hypertension. 2003 Oct;42(4):749-53. doi: 10.1161/01.HYP.0000085220.53285.11. Epub 2003 Jul 21. PMID 12874086
- [Background] Koka V, Huang XR, Chung AC, Wang W, Truong LD, Lan HY. Angiotensin II up-regulates angiotensin I-converting enzyme (ACE), but down-regulates ACE2 via the AT1-ERK/p38 MAP kinase pathway. Am J Pathol. 2008 May;172(5):1174-83. doi: 10.2353/ajpath.2008.070762. Epub 2008 Apr 10. PMID 18403595
- [Background] Dong J, Wong SL, Lau CW, Lee HK, Ng CF, Zhang L, Yao X, Chen ZY, Vanhoutte PM, Huang Y. Calcitriol protects renovascular function in hypertension by down-regulating angiotensin II type 1 receptors and reducing oxidative stress. Eur Heart J. 2012 Dec;33(23):2980-90. doi: 10.1093/eurheartj/ehr459. Epub 2012 Jan 19. PMID 22267242
- [Background] Dai B, David V, Martin A, Huang J, Li H, Jiao Y, Gu W, Quarles LD. A comparative transcriptome analysis identifying FGF23 regulated genes in the kidney of a mouse CKD model. PLoS One. 2012;7(9):e44161. doi: 10.1371/journal.pone.0044161. Epub 2012 Sep 6. PMID 22970174
- [Background] Ejaz AA, Kambhampati G, Ejaz NI, Dass B, Lapsia V, Arif AA, Asmar A, Shimada M, Alsabbagh MM, Aiyer R, Johnson RJ. Post-operative serum uric acid and acute kidney injury. J Nephrol. 2012 Jul-Aug;25(4):497-505. doi: 10.5301/jn.5000173. PMID 22684655
- [Background] el-Agroudy AE, Hassan NA, Foda MA, Ismail AM, el-Sawy EA, Mousa O, Ghoneim MA. Effect of angiotensin II receptor blocker on plasma levels of TGF-beta 1 and interstitial fibrosis in hypertensive kidney transplant patients. Am J Nephrol. 2003 Sep-Oct;23(5):300-6. doi: 10.1159/000072820. Epub 2003 Aug 6. PMID 12904684
- [Background] Haririan A, Metireddy M, Cangro C, Nogueira JM, Rasetto F, Cooper M, Klassen DK, Weir MR. Association of serum uric acid with graft survival after kidney transplantation: a time-varying analysis. Am J Transplant. 2011 Sep;11(9):1943-50. doi: 10.1111/j.1600-6143.2011.03613.x. Epub 2011 Aug 3. PMID 21812917
- [Background] Kanellis J, Watanabe S, Li JH, Kang DH, Li P, Nakagawa T, Wamsley A, Sheikh-Hamad D, Lan HY, Feng L, Johnson RJ. Uric acid stimulates monocyte chemoattractant protein-1 production in vascular smooth muscle cells via mitogen-activated protein kinase and cyclooxygenase-2. Hypertension. 2003 Jun;41(6):1287-93. doi: 10.1161/01.HYP.0000072820.07472.3B. Epub 2003 May 12. PMID 12743010
- [Background] Numakura K, Satoh S, Tsuchiya N, Saito M, Maita S, Obara T, Tsuruta H, Inoue T, Narita S, Horikawa Y, Kagaya H, Miura M, Habuchi T. Hyperuricemia at 1 year after renal transplantation, its prevalence, associated factors, and graft survival. Transplantation. 2012 Jul 27;94(2):145-51. doi: 10.1097/TP.0b013e318254391b. PMID 22728291
- [Background] Feig DI. Hyperuricemia and hypertension. Adv Chronic Kidney Dis. 2012 Nov;19(6):377-85. doi: 10.1053/j.ackd.2012.05.009. PMID 23089272
- [Background] Szabo A, Lutz J, Schleimer K, Antus B, Hamar P, Philipp T, Heemann U. Effect of angiotensin-converting enzyme inhibition on growth factor mRNA in chronic renal allograft rejection in the rat. Kidney Int. 2000 Mar;57(3):982-91. doi: 10.1046/j.1523-1755.2000.00926.x. PMID 10720951
- [Background] Tylicki L, Biedunkiewicz B, Chamienia A, Wojnarowski K, Zdrojewski Z, Aleksandrowicz E, Lysiak-Szydlowska W, Rutkowski B. Renal allograft protection with angiotensin II type 1 receptor antagonists. Am J Transplant. 2007 Jan;7(1):243-8. doi: 10.1111/j.1600-6143.2006.01588.x. PMID 17227571
- [Background] Luque M, Martin P, Martell N, Fernandez C, Brosnihan KB, Ferrario CM. Effects of captopril related to increased levels of prostacyclin and angiotensin-(1-7) in essential hypertension. J Hypertens. 1996 Jun;14(6):799-805. doi: 10.1097/00004872-199606000-00017. PMID 8793704
- [Background] Shah PR, Kute VB, Saboo DS, Goplani KR, Gumber MR, Vanikar AV, Patel HV, Trivedi HL. Safety and efficacy of angiotensin converting enzyme inhibitors and angiotensin receptor blockers in chronic allograft injury. Saudi J Kidney Dis Transpl. 2011 Nov;22(6):1128-32. PMID 22089769
- [Background] Arbeiter K, Pichler A, Stemberger R, Mueller T, Ruffingshofer D, Vargha R, Balzar E, Aufricht C. ACE inhibition in the treatment of children after renal transplantation. Pediatr Nephrol. 2004 Feb;19(2):222-6. doi: 10.1007/s00467-003-1317-8. Epub 2003 Dec 13. PMID 14673630
- [Background] Oudit GY, Herzenberg AM, Kassiri Z, Wong D, Reich H, Khokha R, Crackower MA, Backx PH, Penninger JM, Scholey JW. Loss of angiotensin-converting enzyme-2 leads to the late development of angiotensin II-dependent glomerulosclerosis. Am J Pathol. 2006 Jun;168(6):1808-20. doi: 10.2353/ajpath.2006.051091. PMID 16723697
- [Background] Mizuiri S, Hemmi H, Arita M, Ohashi Y, Tanaka Y, Miyagi M, Sakai K, Ishikawa Y, Shibuya K, Hase H, Aikawa A. Expression of ACE and ACE2 in individuals with diabetic kidney disease and healthy controls. Am J Kidney Dis. 2008 Apr;51(4):613-23. doi: 10.1053/j.ajkd.2007.11.022. Epub 2008 Mar 4. PMID 18371537
- [Background] Mizuiri S, Hemmi H, Arita M, Aoki T, Ohashi Y, Miyagi M, Sakai K, Shibuya K, Hase H, Aikawa A. Increased ACE and decreased ACE2 expression in kidneys from patients with IgA nephropathy. Nephron Clin Pract. 2011;117(1):c57-66. doi: 10.1159/000319648. Epub 2010 Aug 4. PMID 20689326
- [Background] Mizuiri S, Aoki T, Hemmi H, Arita M, Sakai K, Aikawa A. Urinary angiotensin-converting enzyme 2 in patients with CKD. Nephrology (Carlton). 2011 Aug;16(6):567-72. doi: 10.1111/j.1440-1797.2011.01467.x. PMID 21457402
- [Background] Xiao F, Hiremath S, Knoll G, Zimpelmann J, Srivaratharajah K, Jadhav D, Fergusson D, Kennedy CR, Burns KD. Increased urinary angiotensin-converting enzyme 2 in renal transplant patients with diabetes. PLoS One. 2012;7(5):e37649. doi: 10.1371/journal.pone.0037649. Epub 2012 May 22. PMID 22629438
- [Background] Grimm PC, Nickerson P, Gough J, McKenna R, Stern E, Jeffery J, Rush DN. Computerized image analysis of Sirius Red-stained renal allograft biopsies as a surrogate marker to predict long-term allograft function. J Am Soc Nephrol. 2003 Jun;14(6):1662-8. doi: 10.1097/01.asn.0000066143.02832.5e. PMID 12761269

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03317925/Prot_SAP_000.pdf